CLINICAL TRIAL: NCT02461316
Title: Open, Non-Interventional, Multicentre Trial of Rituximab in Combination With FC for the First-Line Therapy of Patients With Chronic Lymphocytic Leukaemia
Brief Title: Rituximab in Combination With Fludarabine and Cyclophosphamide in Patients With Chronic Lymphocytic Leukemia
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML25066
Record Dates: First submitted 2015-06-01; First posted 2015-06-03 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Lymphocytic Leukemia, Chronic, Chronic Lymphocytic Leukemia, Cancer
MeSH Terms: conditions — Leukemia, Lymphoid; Bronchiolitis Obliterans Syndrome; Leukemia, Lymphocytic, Chronic, B-Cell; Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Combination Treatment in Chronic Lymphocytic Leukemia (CLL): All participants receiving combination treatment in Chronic Lymphocytic Leukemia (CLL)
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention administered in this study: Rituximab in combination with fludarabine and cyclophosphamide for 6 months according to registered indication.

SUMMARY:
Evaluation of safety profile and tolerability of MabThera (rituximab) in combination with chemotherapy (fludarabine and cyclophosphamide) in the treatment of Chronic Lymphocytic Leukemia (CLL).

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years with diagnosed Chronic Lymphocytic Leukemia (CLL)
* CLL stages: Binet stage C (Rai III or IV), Binet stage B (Rai I and II) requiring treatment

Exclusion Criteria:

- Patients who are not eligible for rituximab treatment according to Summary of Product Characteristics (SmPC)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Previously untreated patients with Chronic Lymphocytic Leukemia (CLL)
Sampling Method: Non-Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2009-07; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Percentage of Adverse Events (AEs) | From baseline to end of study up to 18 months
Percentage of Serious Adverse Events (SAEs) | From baseline to end of study up to 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (3):
- Serbia (3):
  - Belgrade
  - Kragujevac
  - Novi Sad